CLINICAL TRIAL: NCT00814983
Title: Myeloablative Allogeneic Stem Cell Transplantation Using a Naive T-Cell Depleted Peripheral Blood Stem Cell Graft
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: IND approval for naive T-cell depletion not obtained
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000993
Record Dates: First submitted 2008-12-26; First posted 2008-12-29 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-09

CONDITIONS: ALL; ANLL; MDS; NHL
Keywords: myeloablative; stem cell; naive T-cell depleted; allogeneic
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naive T-cell Depleted Stem Cell Transplant (Experimental): Experimental: Cohort 2 will receive a T-cell depleted peripheral blood stem cell graft. All other aspects of this stem cell transplantation are in line with the standard of care.
  Interventions: Procedure: Naive T-cell Depleted Stem Cell Transplant; Device: Isolex device from Baxter
- Stem Cell Transplant No Manipulation (Active Comparator): Control: Cohort 1 Stem Cell Transplant No Manipulation will receive the currently accepted standard approach to myeloablative allogeneic stem cell transplantation
  Interventions: Procedure: Stem Cell Transplant No Manipulation

INTERVENTIONS:
Procedure: Naive T-cell Depleted Stem Cell Transplant — The Isolex device from Baxter will be used to perform the cell selection procedure. After the CD34 selected stem cell graft has been collected, the CD34- "flow-through"fraction will be depleted of CD45RA+ naive T-cells. To accomplish this, a second immunomagnetic bead selection process will be performed on the Isolex device, making use of a GMP-grade murine anti-human CE45RA antibody. This depleted fraction will comprise the donor lymphocyte inoculum given to the transplant recipient along with the stem cell component on day 0 of transplant.
  Arms: Naive T-cell Depleted Stem Cell Transplant
Procedure: Stem Cell Transplant No Manipulation — These patients will be transplanted with unmanipulated peripheral blood stem cells.
  Arms: Stem Cell Transplant No Manipulation
Device: Isolex device from Baxter
  Arms: Naive T-cell Depleted Stem Cell Transplant

SUMMARY:
The primary objectives will be to measure the safety and efficacy of allogeneic stem cell transplantation using a peripheral blood stem cell graft that has been depleted of CD45RA+ Naive T-cells.

The secondary objectives will be to measure the pace of immune recovery.

DETAILED DESCRIPTION:
A cohort of patients (Cohort 1) will be enrolled to receive the currently accepted standard approach to myeloablative allogeneic stem cell transplantation. With the exception of volume and/or plasma depletion (in cases of donor/recipient ABO incompatibility), the peripheral blood stem cell graft will be unmodified. The primary purpose of Cohort 1 is to prospectively collect samples for measurement of immune recovery from a relatively homogeneous population of patients treated in a uniform manner. Within the limitations of age-matching, patients accrued to Cohort 1 will be incorporated into a larger retrospective historical control group for purposes of comparison with Cohort 2 of the incidence of grade II-IV acute Graft versus Host disease. The experimental aspects of this trial will be the use of a naïve T-cell depleted peripheral blood stem cell graft (Cohort 2). All other aspects of this stem cell transplantation are in line with the standard of care. Recruitment to this trial will be stratified by donor type as matched sibling or matched unrelated donor. Patients will be conditioned with total body irradiation (1350cGy) and Cyclophosphamide. The donor stem cell grafts will come from mobilized peripheral blood of 6/6 HLA-identical family members or 8/8 (HLA A, B, C, DRB1) allele-level matched unrelated donors.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years.
* 8/8 or 7/8 HLA-identical matched sibling OR Allele level 8/8 (HLA-A, B, C, DRbeta1) matched unrelated donor.
* Patients with high risk ALL in first complete remission, with high risk being defined by the presence of t(4;11), t(9;22) or t(1;19) or patients presenting with extreme hyperleukocytosis (WBC>500,000/ml) or partial remission after initial induction therapy.
* Adult patients with acute non-lymphocytic Leukemia (ANLL) in first complete remission with high-risk cytogenetics (monosomy chromosome 5 or 7, del(5q), abn(3q26), complex karyotypic abnormalities) or failure to achieve complete remission after standard induction therapy.
* All patients with ALL or ANLL in second or subsequent remission or partial remission (<5% blasts in bone marrow as measured by flow cytometry).
* All patients with CML in chronic (failed interferon and/or Gleevec) or accelerated phase.
* Patients with myelodysplastic syndrome with International Prognostic Scoring System (IPSS) risk category of INT-1 or greater.
* Myelofibrosis with myeloid metaplasia
* Patients with severe aplastic anemia must have failed immunosuppressive therapy such as cyclosporine plus anti-thymocyte globulin.
* Patients with a history of CNS disease must have been treated and have no active CNS disease at the time of protocol treatment.
* ECOG performance status <2
* Patients must have adequate function of other organ systems as measured by:
* Creatinine clearance (by Cockcroft Gault equation [Appendix IV]) > 30ml/min. Hepatic transaminases (ALT/AST) < 4 x normal, bilirubin < 2.0 mg/dl.
* Pulmonary function tests demonstrating FVC and FEV1 of >50% of predicted for age and DLCO > 50% of predicted.
* Ejection fraction of >45% by echocardiogram, radionuclide scan or cardiac MRI.
* Patients must be HIV negative.
* Patients must not be pregnant.

Exclusion Criteria:

* Patients with > 5% blasts in bone marrow or peripheral circulation.
* Patients with rapidly progressive ANLL or ALL.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Horwitz, MD, Principal Investigator — Duke Health

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stem Cell Transplant No Manipulation | Naive T-cell Depleted Stem Cell Transplant
Started | 15 | 0
Completed | 12 | 0
Not Completed | 3 | 0
Not completed — Screen failure | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Graft failure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stem Cell Transplant No Manipulation | Naive T-cell Depleted Stem Cell Transplant | Total
Number analyzed (Participants) | 15 | 0 | 15
Age Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 15 |  | 15
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 8 |  | 8
  Male | 7 |  | 7
Region of Enrollment [Number; unit: participants]
  United States | 15 |  | 15

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Grade II-IV Acute Graft Versus Host Disease
Time Frame: One year from date of transplant
Population: No analysis was performed since the experimental arm was not opened
Arm/Group | Stem Cell Transplant No Manipulation | Naive T-cell Depleted Stem Cell Transplant
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Disease Free Survival
Time Frame: One year
Population: No analysis was performed since the experimental arm was not opened
Arm/Group | Stem Cell Transplant No Manipulation | Naive T-cell Depleted Stem Cell Transplant
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Rate of Immune Recovery
Description: The time to recovery of T-cell subset, B cell and NK cell recovery will be monitored along with T-Cell proliferative response to mitogens.
Time Frame: 3 years
Population: No analysis was performed since the experimental arm was not opened
Arm/Group | Stem Cell Transplant No Manipulation | Naive T-cell Depleted Stem Cell Transplant
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event analysis was not undertaken due to stopping the study prior to enrolling in the experimental arm.
Arm/Group | Stem Cell Transplant No Manipulation | Naive T-cell Depleted Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes